CLINICAL TRIAL: NCT04870424
Title: Colchicine for Patients With Aortic Stenosis Undergoing Transcatheter Aortic Valve Replacement (Co-STAR): a Randomized-controlled Trial
Brief Title: Colchicine for Patients With Aortic Stenosis Undergoing Transcatheter Aortic Valve Replacement
Acronym: Co-STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Co-STAR
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Transcatheter Aortic Valve Replacement; Atrial Fibrillation New Onset; Pacemaker; Colchicine
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental)
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine in a loading dosage of 1mg single dose per os the day before TAVI and 1mg single dose at the day of procedure. Thereafter, colchicine 0.5mg once daily per os up to post-procedural day 12.
  Arms: Colchicine
Drug: Placebo — Placebo once daily per os the day before TAVI and once at the day of procedure. Thereafter, once daily per os up to post-procedural day 12.
  Arms: Placebo

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a well-established alternative to surgical aortic valve replacement for the treatment of patients with symptomatic severe aortic stenosis. While peri-procedural complications such as stroke, vascular complications and bleeding have substantially declined with the refinement of transcatheter valves and increasing experience, new-onset atrial fibrillation (NOAF) or atrioventricular conduction disturbances continue to occur in almost half of all patients.

Colchicine is a well-known substance that has been approved for the treatment of acute gout flares and familial Mediterranean fever in many countries. Colchicine has proven safe and effective in the prevention of atrial fibrillation after cardiac surgery. The anti-inflammatory effects of colchicine may mitigate the occurrence of atrioventricular conduction disturbances and thus the need for the implantation of a permanent pacemaker post transcatheter aortic valve implantation.

The objective of the Co-STAR-Trial is to investigate the efficacy of colchicine for the prevention of new-onset atrial fibrillation and conduction disturbances requiring the implantation of a permanent pacemaker in patients undergoing transcatheter aortic valve implantation.

Co-STAR is an investigator-initiated, randomized, double blind, placebo-controlled trial. A total of 200 patients referred for treatment of symptomatic severe aortic stenosis and selected to undergo TAVI will be randomized in a 1:1 ratio to the treatment with Colchicine or placebo for 30 days post transcatheter aortic valve implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. Symptomatic severe aortic stenosis defined by an aortic valve area (AVA) ≤1.0 cm2 or an AVA indexed to body surface area <0.6cm2/m2
3. Selected to undergo transfemoral TAVI based on heart team decision

Exclusion Criteria:

1. Life expectancy <1 year irrespective of valvular heart disease
2. Kidney disease with a creatinine clearance ≤30 ml/min
3. Known severe liver disease
4. Known neuromuscular disease
5. Clinically significant anaemia with haemoglobin <80g/L
6. Known inflammatory bowel disease or chronic diarrhea
7. Known ongoing bacterial infection
8. Known galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
9. Current treatment with colchicine, steroids or biologicals for any indication
10. Concomitant intake of Cyclosporine, Amiodarone, Clarithromycin, Erythromycin, Omeprazole, Verapamil or other strong inhibitors of CYP3A4 or P-Glycoprotein
11. Concomitant intake of Carbamazepin, Phenobarbital, Phenytoin, Rifampicin or other strong inductors of CYP3A4 and P-Glycoprotein
12. Permanent pacemaker or implantable cardioverter defibrillator
13. History of atrial fibrillation
14. Absence of sinus rhythm on hospital admission
15. Planned non-cardiac surgery within 30 days
16. Known intolerance to colchicine
17. Inability to provide written informed consent
18. Known or suspected non-compliance, drug or alcohol abuse
19. Participation in another clinical trial with an active intervention
20. Any other planned cardiac intervention performed in the 7 days before TAVI, concomitantly with TAVI or in the 30 days after TAVI except for percutaneous coronary interventions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of the composite of new onset atrial fibrillation or occurrence of conduction disturbances requiring the implantation of a permanent pacemaker | 30 days
  Assessed based on extended rhythm monitoring performed until 7 days post-discharge as well as clinically or incidentally captured episodes of NOAF captured during routine care thereafter. NOAF is defined as at least one episode of atrial fibrillation with a duration >30s.

SECONDARY OUTCOMES:
Single components of primary composite endpoint | 30 days and 1 year
  Including predefine sensitivity analysis using the alternative definition of NOAF: At least one episode of atrial fibrillation with a duration >6 min.
The incidence of conductance disturbances | 30 days, 1 year
  New or worsened first-degree atrioventricular (AV) block, second-degree AV block (Mobitz I or Mobitz II), high-grade atrioventricular block, third-degree AV block, right bundle branch block, left bundle branch block, left anterior fascicular block, left posterior fascicular block, intraventricular conduction delay
The predictors of conductance disturbances | 30 days, 1 year
  New or worsened first-degree atrioventricular (AV) block, second-degree AV block (Mobitz I or Mobitz II), high-grade atrioventricular block, third-degree AV block, right bundle branch block, left bundle branch block, left anterior fascicular block, left posterior fascicular block, intraventricular conduction delay
The incidence of new arrhythmias resulting in hemodynamic instability or requiring therapy | 30 days, 1 year
  Defined as electrical/medical cardioversion or initiation of a new medication e.g. oral anticoagulation, rhythm, or rate controlling therapy
Inflammatory marker levels | at day 1
  IL-6, IL-8, TNF-alpha, IL-1β, CRP, high-sensitivity CRP
The proportion of patients with at least one prosthetic leaflet with > 50% motion reduction or with at least one prosthetic leaflet with thickening | 30 days
  Based on a study-specific cardiac computed tomography angiography
The proportion of prosthetic leaflets with > 50% motion reduction or leaflet thickening | 30 days
  Based on a study-specific cardiac computed tomography angiography
The incidences of major clinical adverse events | 30 days, 1 year
  All-cause mortality, stroke, systemic embolism, myocardial infarction, infections, clinical valve thrombosis

OTHER OUTCOMES:
Safety Outcome | 30 days
  Incidence of gastrointestinal side effects and clinically severe side effects possibly related to study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Prof., Principal Investigator — University of Bern, Switzerland
Locations (1):
- Inselspital, Bern University Hospital, Department of Cardiology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryffel C, Lanz J, Guntli N, Samim D, Furholz M, Stortecky S, Tomii D, Heg D, Boscolo Berto M, Peters AA, Reineke D, Reichlin T, Grani C, Windecker S, Pilgrim T. Colchicine in patients with aortic stenosis undergoing transcatheter aortic valve replacement: a double-blind randomized trial. Nat Commun. 2025 Jul 15;16(1):6501. doi: 10.1038/s41467-025-61916-6. PMID 40659682